CLINICAL TRIAL: NCT02031952
Title: Hepatectomy Versus Hepatectomy With Lymphadenectomy in Hepatocellular Carcinoma ----A Prospective Randomized Controlled Clinical Trail
Brief Title: Hepatectomy Versus Hepatectomy With Lymphadenectomy in Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rvrl2005
Record Dates: First submitted 2014-01-04; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; hepatectomy; lymphadenectomy; complication; prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Lymph Node Excision; Hepatectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hepatectomy combined lymphadenectomy (Experimental): hepatectomy combined lymphadenectomy
  Interventions: Procedure: hepatectomy combined with lymphadenectomy
- hepatectomy (Active Comparator): hepatectomy alone
  Interventions: Procedure: hepatectomy alone

INTERVENTIONS:
Procedure: hepatectomy combined with lymphadenectomy
  Arms: hepatectomy combined lymphadenectomy
Procedure: hepatectomy alone
  Arms: hepatectomy

SUMMARY:
The preventive lymphadenectomy is not performed routinely for hepatocellular carcinoma (HCC) patients in clinical practice. While many patients suffered the recurrence without the evidence of portal or hepatic vascular invasion or multiple loci, it lead to reconsider the value of preventive resection of regional lymph node for those patients. Recently, more and more studies had found the incidence of lymph node metastasis was higher in autopsy specimen than those in operable patients.

This project is a prospective randomized controlled trial, planning to compare hepatectomy with hepatectomy combined lymphadenectomy regarding of the safety and efficacy in HCC patients, to reach a further understanding of the role of lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years;
* Eastern Cooperative Oncology Group (ECOG) Performance Status is grade 0 or 1;
* good liver function with Pugh-Child Class A or B;
* indocyanine green retention at 15 minutes (ICG-R15) <15%;
* without severe cirrhosis;
* the diameter of tumor is equal to or more than 3 cm;
* the liver resection could be assessed R0 (the define of R0 resection will be explained in the section of Surgical procedures);
* absence of extrahepatic metastasis.

Exclusion Criteria:

* the diameter of tumor is less than 3 cm;
* palliative resection of tumor;
* with the history of hepatic encephalopathy, ascites, and variceal bleeding;
* with severe hepatic cirrhosis;
* tumor rupture;
* with the history of upper abdominal surgery, it is tough to remove the regional lymph nodes; or it is unable to be resected when multiple lymph nodes mixed and fixed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival | 5 year
  The recurrence-free survival time was defined as the time from the date of resection or ablation to the time of recurrence, metastasis or last follow-up.

SECONDARY OUTCOMES:
Post-operation complication | 90-d after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Yuan, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China